CLINICAL TRIAL: NCT03064607
Title: Measurement of Biomarkers of Neurodegeneration in Newborns After Exposure to Anesthetics
Brief Title: Neurodegeneration in Newborns After Anesthetics
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 812651
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Neurodegeneration; General Anesthesia
Keywords: Neonates; biomarkers; EXIT procedure; Cesarean Section
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: Women undergoing c-section or EXIT procedure
  Interventions: Other: Fluid collection

INTERVENTIONS:
Other: Fluid collection — Fluids tested for biomarker S100beta

SUMMARY:
The purpose of the study is to quantify biomarkers of neural damage in neonates exposed to varying levels of volatile anesthetic in utero.

DETAILED DESCRIPTION:
This study will enroll 130 pregnant patients undergoing C-section or fetal surgery with EXIT (Ex Utero Intrapartum Treatment) procedures under epidural or general anesthesia with low (0.75 MAC) or high (2.5 MAC) concentrations of desflurane. Patients will be recruited from both the Hospital of the University of Pennsylvania (100 C Section) and Children's Hospital of Philadelphia (30 EXIT procedure).

The standard of care protocol for patients undergoing anesthesia for these cases will be followed throughout the surgery. These include monitoring and management of blood pressure, heart rate and rhythm, ventilation, oxygenation, temperature, and fluid status. Management of these parameters will be at the discretion of the clinical team. The choice of the anesthetic technique will also be at the discretion of the clinical team. Typical anesthetic management includes the following:

C-section under epidural anesthesia: induction and maintenance with 1.5% lidocaine, sodium bicarbonate and 1:200,000 epinephrine

C-section under general anesthesia: induction with propofol 2 mg/kg and succinylcholine 2 mg/kg intravenously; maintenance with desflurane 4.5-5%

EXIT procedure under general anesthesia: induction with propofol 2 mg/kg and succinylcholine 2 mg/kg intravenously; maintenance with desflurane 15-18%

1. After the baby is delivered, and the umbilicus is cut, two ml of blood will be taken from the umbilical vein and artery on the placenta side. A portion of the blood will be used for the blood gas and the remainder will be used for the S100B study assay.
2. 5 ml of blood will be taken from the mother via the existing intravenous catheter.
3. 5 ml of amniotic fluid will be obtained at hysterotomy and will be used for the S100B study assay.

All subjects will receive standard of care post operative clinical care and monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Women delivering a child via cesarean section or EXIT procedure
2. Informed consent

Exclusion Criteria:

1. Known fetal neurologic defect
2. Known maternal neurologic abnormality
3. Sensitivity or allergy to medications used in the study

   1. C-section under epidural anesthesia: induction and maintenance with 1.5% lidocaine, sodium bicarbonate and 1:200,000 epinephrine
   2. C-section under general anesthesia: induction with propofol 2 mg/kg and succinylcholine 2 mg/kg intravenously; maintenance with desflurane 4.5-5%
   3. EXIT procedure under general anesthesia: induction with propofol 2 mg/kg and succinylcholine 2 mg/kg intravenously; maintenance with desflurane 15-18%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-11-05 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
S100β Umbilical | 1 day
  as measured by the concentration of biomarker in umbilical arterial and venous blood

SECONDARY OUTCOMES:
S100β Amniotic | 1 day
  as measured by the concentration of biomarker in maternal amniotic fluid
S100β Blood | 1 day
  as measured by the concentration of biomarker in maternal blood
Blood gas | 1 day
  as measured by the results of umbilical arterial and venous blood

CONTACTS AND LOCATIONS:
Overall Officials: Huafeng Wei, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No